CLINICAL TRIAL: NCT06631313
Title: A Prospective, Uncontrolled, Open-label Healthy Volunteer Study to Assess the Performance of the PureWick™ Male and PureWick™ Flex Female External Catheter Devices in Adolescents
Brief Title: PureWick™ Adolescent Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UCC-23AC023
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers, Adolescent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PureWick System (Experimental)
  Interventions: Device: PureWick System

INTERVENTIONS:
Device: PureWick System — The PureWick System consists of the PureWick Urine Collection System used with either the PureWick Male External Catheter or the PureWick Flex Female External Catheter, which are intended for non-invasive urine output management.

SUMMARY:
A prospective, uncontrolled, open-label healthy volunteer study to assess the performance of the PureWick Male and PureWick Flex Female external catheter devices in adolescents

DETAILED DESCRIPTION:
The objective of this healthy volunteer study is to understand if external catheters are an effective alternative in the adolescent population in both male and female adolescents. The main question it aims to answer is: Do the PureWick Male and PureWick Flex female external catheters effectively capture urine in the adolescent population after both healthcare professional placement and self-placement? Participants will void while wearing the external catheter two times and answer brief questionnaires assessing perceived wetness, IFU comprehension, comfort and ease of use. Total study participation time is 2-3 hours in a single day.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Adolescent Male or Female aged 12 through 21 years old
2. Able to independently and voluntarily void urine
3. Ability to speak and understand English.
4. Willing to comply with all study procedures in the protocol.
5. Provision of signed and dated informed consent form.

Exclusion Criteria:

1. Has urinary retention
2. Incontinent to feces
3. Has any irritation, wound, open lesion at the device application site.
4. For females: currently menstruating without use of an internal device, e.g. tampon or menstrual cup, during the execution of the study.
5. For females: currently pregnant at time of consenting (self-reported)
6. Currently enrolled in or has previously been enrolled in or has completed nursing or other clinical training and courses.
7. Has ever been employed as a home health aide or homecare provider.
8. Any other condition that, in the opinion of the investigator, would preclude them from participating in the study.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2024-08-28 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- TKL Research, Inc., Fair Lawn, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PureWick System
Started | 43
Female Participants | 20
Male Participants | 23
Healthcare Professional Placed Device | 42
Self-Placed Device | 42
Completed | 41
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | PureWick System
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.8 (2.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 21
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43
BMI [Mean (Standard Deviation); unit: kg/m2] | 25.37 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Performance of the PureWick System in Adolescents After HCP Placement and Self-placement
Description: Capture rate following void (captured as % of urine captured by device and collected in canister, measured by weight).
  Prior to each void, the weight of the empty urine collection canister and the weight of a dry absorbent pad are collected. Participants void into the device while laying in a bed with the absorbent pad underneath them. After each void, the post-void weight of the urine collection canister and the post-void weight of the absorbent pad are collected.
  Capture rate is calculated as the weight of captured urine (post-void canister weight - pre-void canister weight) / total urine volume (captured urine (post-void canister weight - pre-void canister weight) + leaked urine (post-void pad weight - pre-void pad weight)) * 100.
Time Frame: Approximately 2 hours after device placement
Population: All evaluable participants defined as those who voided with the device in place.
Measure: Mean (Standard Deviation); unit: Percentage of urine captured
Groups:
- Healthcare Professional Placed Device: Evaluation of the PureWick System after being placed on the participant by a healthcare professional (HCP).
- Self-Placed Device: Evaluation of the PureWick System after being self-placed by the participant.
Arm/Group | Healthcare Professional Placed Device | Self-Placed Device
Number analyzed (Participants) | 41 | 41
Percentage of urine captured
  Overall (Females & Males Combined) | 90.40 (19.31) | 93.09 (13.79)
  PureWick Flex Female: number analyzed (Participants) | 18 | 18
  PureWick Flex Female | 87.15 (17.43) | 90.41 (7.91)
  PureWick Male: number analyzed (Participants) | 23 | 23
  PureWick Male | 92.95 (20.69) | 95.19 (16.95)

2. Secondary Outcome: Participant Comfort
Description: Overall comfort on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Uncomfortable, 2 = Uncomfortable, 3 = Neither Comfortable or Uncomfortable, 4 = Comfortable, and 5 = Very Comfortable.
  The last survey question related to likelihood to recommend the device ranged from 1-5 with higher scores indicating a better outcome, where 1 = Very Unlikely, 2 = Unlikely, 3 = Neither Likely Nor Unlikely, 4 - Likely, and 5 = Very Likely.
Time Frame: Approximately 2 hours after device placement
Population: All enrolled participants that completed a comfort questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PureWick Flex Female: PureWick Flex Female External Catheter, which is intended for non-invasive urine output management.
- PureWick Male: PureWick Male External Catheter, which is intended for non-invasive urine output management.
Arm/Group | PureWick Flex Female | PureWick Male
Number analyzed (Participants) | 18 | 23
score on a scale
  Device Placement Comfort | 4.4 (0.61) | 4.3 (0.82)
  Device Voiding Comfort | 4.2 (0.81) | 4.3 (0.76)
  Device Removal Comfort | 4.7 (0.46) | 4.0 (1.02)
  Likelihood to Recommend Device to a Loved One | 4.3 (0.69) | 4.1 (1.06)

3. Secondary Outcome: Participant Ease of Use
Description: Ease of use score on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Difficult, 2 = Somewhat Difficult, 3 = Average Difficulty, 4 = Somewhat Easy
Time Frame: Approximately 2 hours after device placement
Population: All enrolled participants that completed an ease-of-use questionnaire after device self-placement.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Flex Female | PureWick Male
Number analyzed (Participants) | 19 | 23
score on a scale
  Ease of Use during Device Placement | 4.4 (0.78) | 4.3 (0.69)
  Ease of Use during Device Removal | 5.0 (0.00) | 4.7 (0.65)

4. Secondary Outcome: IFU Comprehension
Description: Overall IFU comprehension on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Strongly Disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, and 5 = Strongly Agree.
Time Frame: Approximately 2 hours after device placement
Population: All enrolled participants that completed an IFU Comprehension questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Flex Female | PureWick Male
Number analyzed (Participants) | 18 | 23
score on a scale
  I was able to understand and follow the written instructions | 4.8 (0.43) | 4.7 (0.56)
  I was able to understand the pictures in the instructions | 4.8 (0.38) | 4.7 (0.45)
  I was able to place the PureWick device on myself | 4.7 (0.46) | 4.6 (0.66)

5. Secondary Outcome: HCP Ease of Use
Description: Ease of use score on a 5-point Likert scale ranging from 1- 5 with higher scores indicating a better outcome, where 1 = Very Difficult, 2 = Somewhat Difficult, 3 = Average Difficulty, 4 = Somewhat Easy, and 5 = Very Easy.
Time Frame: From date of first enrollment until the date of last patient completion, approximately 4 weeks
Population: All HCPs who completed an ease-of-use questionnaire after placing at least one device on study participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PureWick Flex Female | PureWick Male
Number analyzed (Participants) | 3 | 5
score on a scale
  Ease of Use during Device Placement | 5.0 (0.00) | 5.0 (0.00)
  Ease of Use during Device Removal | 5.0 (0.00) | 5.0 (0.00)

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | PureWick System
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT06631313/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT06631313/SAP_001.pdf